CLINICAL TRIAL: NCT02349204
Title: The Effect of Music on Surgical Skill in the Setting of Simulated Intraocular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015-1938
Record Dates: First submitted 2015-01-05; First posted 2015-01-28 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Surgical Performance
Keywords: Simulator; Music; Mozart Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure to music (Experimental): The participants in this groups will have to complete the tasks on the intraocular surgery simulator while listening to Mozart's sonata for 2 pianos in D-440
  Interventions: Behavioral: Music - Mozart's sonata for 2 pianos in D-440
- No exposure (No Intervention): The participants in this groups will have to complete the tasks on the intraocular surgery simulator in silence

INTERVENTIONS:
Behavioral: Music - Mozart's sonata for 2 pianos in D-440
  Arms: Exposure to music

SUMMARY:
Music is commonly heard in operating room. The goal of this study is to measure the effect of music on surgical performance using a intraocular surgery simulator. The music chosen is Sonata for 2 pianos D-440 from Mozart. The participants will complete 2 tasks on the simulator, both with and without music, in a randomized sequence. The results will be subtracted from the simulator and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ophthalmology residents at Laval University
* Ophthalmologist at Centre Hospitalier Universitaire de Québec

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Task score | Assessed up to 12 weeks after randomization
  The participants will perform tasks on a simulator on three separate days. The outcome will be measured at each of these visits.

SECONDARY OUTCOMES:
Time to complete the task | Assessed up to 12 weeks after randomization
  The participants will perform tasks on a simulator on three separate days. The outcome will be measured at each of these visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Caissie, MD, FRCPC, Principal Investigator — Centre de recherche du CHU de Québec : Université Laval
Locations (1):
- Centre Universitaire d'Ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Canada